CLINICAL TRIAL: NCT05298878
Title: Virtual Physical Rehabilitation for Patients Living with Long COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); RESPIPLUS (Unknown); Santé WillKin (WillKin Health) (Unknown); Canadian Thoracic Society (Unknown)
Responsible Party: Principal Investigator, Tania Janaudis-Ferreira, Scientist, Translational Research in Respiratory Diseases Program, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-8559
Record Dates: First submitted 2022-03-24; First posted 2022-03-28 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; Post COVID-19; Long COVID
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual home-based rehabilitation plus usual outpatient care (Experimental): An 8-week home-based virtual rehabilitation program consisting of exercises and education plus usual care.
  Interventions: Other: Intervention Group: Virtual home-based rehabilitation plus usual outpatient care
- Usual outpatient care (No Intervention): The control group will receive usual outpatient care which consists of any medical outpatient follow-up visits. The participants will receive a set of written generic instructions on how to manage symptoms and engage in physical activity after critical illness.

INTERVENTIONS:
Other: Intervention Group: Virtual home-based rehabilitation plus usual outpatient care — 14 supervised exercise virtual sessions with Kinesiologist and 10 independent exercise sessions. Each session lasts 40 minutes. The exercises consist of aerobic training; functional lower and upper body strengthening; balance; and flexibility exercises. During the first 10 minutes of the first session of each week, there is an educational session.
  Week 1-2: three supervised virtual sessions Week 3-4: two supervised virtual sessions and one independent session. Week 5-8: one supervised virtual session and two independent sessions.
  Arms: Virtual home-based rehabilitation plus usual outpatient care

SUMMARY:
The purpose of this study is to investigate whether a timely, virtual home-based physical rehabilitation program for patients living with long COVID can improve functional mobility compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

(i) adult patients (18+ years old) who have had a confirmed or probable COVID-19 infection and who have self-reported persisting symptoms of either reduced mobility, muscle weakness, dyspnea, or fatigue;

(ii) participants must be technologically capable of connecting (either independently or through household members) with an online videoconferencing platform through an e-mail invitation; and

(iii) be able to collaborate with the research assistant to complete the virtual assessment sessions or have a family member available to help.

Exclusion Criteria:

(i) pre-existing or newly identified severe cognitive impairment;

(ii) inability to speak or comprehend English or French;

(iii) known or self-reported acute and/or uncontrolled cardiac, musculoskeletal, or neurological condition that might render rehabilitation participation unsafe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Change in the basic mobility domain of the Activity Measure for Post-Acute Care (AM-PAC) | Baseline, Week 8 (up to 1 week), and at 6 months.
  The AM-PAC is a validated, self-reported instrument assessing activity limitations based on the International Classification of Functioning, Disability, and Health (ICF). Each item is scored from 1 (unable to perform) to 4 (none or no difficulty) with lower scores indicating lower levels of function.

SECONDARY OUTCOMES:
Change in lower-body strength | Baseline, Week 8 (up to 1 week), and at 6 months.
  The 1-minute sit-to-stand test (1-min STS) is feasible to use in hospital survivors of COVID-19. It is used to assess lower body-strength, exercise tolerance, and exertional desaturation. The score is the total number of stands within one minute.
Change in functional mobility | Baseline, Week 8 (up to 1 week), and at 6 months.
  The fast-Timed-Up-and-Go test (TUG) assesses physical function and functional mobility. The score consists of the time taken to complete the test activity, in seconds.
Change in fatigue | Baseline, Week 8 (up to 1 week), and at 6 months.
  Measured by the Fatigue Visual Analog Scale.
Change in dyspnea | Baseline, Week 8 (up to 1 week), and at 6 months.
  Measured by the Transition Dyspnea Index.
Change in health-related quality of life | Baseline, Week 8 (up to 1 week), and at 6 months.
  Measured by the Short Form 12-item Health Survey (SF-12).
Change in health state utilities | Baseline, Week 8 (up to 1 week), and at 6 months.
  Measured by the EuroQol 5-dimension 5-level Questionnaire (EQ-5D-5L).
Change in anxiety and depression | Baseline, Week 8 (up to 1 week), and at 6 months.
  Measured by the Hospital Anxiety and Depression Scale.
Change in cognitive function | Baseline, Week 8 (up to 1 week), and at 6 months.
  Measured by the AM-PAC Cognition Subscale.
Change in the degree of distress in response to trauma | Baseline, Week 8 (up to 1 week), and at 6 months.
  Measured by the Impact of Event Scale - Revised.
Self-reported health service use | 30 days after the 8-week period.
  Doctors visits, emergency department visits and hospital readmission etc.

CONTACTS AND LOCATIONS:
Overall Officials: Tania Janaudis-Ferreira, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Marla Beauchamp, PDF, Principal Investigator — McMaster University; Jean Bourbeau, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - McMaster University, Hamilton, Ontario
  - Research Institute, McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Summary results will be available on the trial registry site within 12 months from the last visit of the last participant.
  Other data will be shared on request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 12 months from the last visit of the last participant.
Access Criteria: Access to anonymized IPD can be requested by researchers.